CLINICAL TRIAL: NCT02377544
Title: The Role of Bifidobacterium Animalis Ssp Lactis DR10 Supplementation in Women During Pregnancy and Lactation on Breast Milk IL-8 and Gut Mucosa Integrity in Infant
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Naomi Esthernita (Other)
Responsible Party: Sponsor-Investigator, Naomi Esthernita, MD, Indonesia University
Organization: Indonesia University (Other)
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: FKUI-RSCM
Record Dates: First submitted 2015-02-26; First posted 2015-03-03 (Estimated); Last update posted 2016-02-25 (Estimated); Status verified 2016-02

CONDITIONS: Bifidobacterium
MeSH Terms: interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Saccharum lactis
  Interventions: Other: Placebo
- Probiotic (Experimental): Bifidobacterium animalis lactis
  Interventions: Dietary Supplement: Probiotic

INTERVENTIONS:
Dietary Supplement: Probiotic
  Arms: Probiotic
Other: Placebo
  Arms: Placebo

SUMMARY:
Hopefully this research can help to provide the optimal nutrition management from pregnancy so that the babies wiil born with better quality of health and reduce the morbidity and mortality.

Until now, there is no data regarding probiotics in Indonesien breastmilk and the role of probiotics supplementation on pregnant women to the baby especially from inflammation pathways. The investigators hope the result of this research can help reducing infant morbidity and mortality rate in Indonesia, also has a benefit for future research.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women ,gestation age 32-34 weeks, normal pregnancy, plan to deliver spontaneously, no antibiotic
* tend to give exclusive breastfeeding
* want to join the research
* well doing baby

Exclusion Criteria:

* pregnant women with pre-eclampsia,bleeding,infection,premature rupture of the membrane or other chronic disease
* plan to deliver by caesarean section

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2014-12; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Gastrointestinal microbiota examination by DNA extraction and real time PCR | 3 months
Examination of IL-8 in breast milk | 3 months
Examination of urine IFABP | 3 months
Calprotectin examination in stool of infants aged 3 months | 3 months
Alpha 1 antitrypsin | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Budi Kemuliaan Women and Children Hospital, Jakarta, Central Jakarta, Indonesia